CLINICAL TRIAL: NCT02829047
Title: A Prospective, Multicenter, Open-label, Single-arm Study to Assess the Tolerability, Safety and Efficacy of a New Frequency of Vibrant Capsule Administration
Brief Title: Tolerability, Safety and Efficacy of a New Frequency of Vibrant Capsule Administration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted at interim analysis to allow the sponsor to focus on a new study with different design.
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 220CLD
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2017-03

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vibrating Capsule (Other): Patients will receive vibrating capsule for 6 weeks of treatment (14 capsules in 3 weeks)
  Interventions: Device: Vibrating Capsule

INTERVENTIONS:
Device: Vibrating Capsule — Patients will receive vibrating capsule for 6 weeks of treatment (14 capsules in 3 weeks)

SUMMARY:
The study is a prospective, multicenter, open-label, single-arm study, to evaluate the tolerability, safety and efficacy of the Vibrant Capsule in relieving constipation.

DETAILED DESCRIPTION:
One arm will be assessed: Vibrant Capsule administered with a sequence of one per day for 2 days, followed by one day without, one per day for 2 days followed by one day without, etc. (14 capsules in 3 weeks).

The study will have one interim analysis.

Patients will follow a 2 weeks baseline period and then take the Vibrant Capsule for a treatment period of 6 weeks.

Data reporting will be done on an electronic Case Report Form and an eDiary. During the 2 weeks of baseline, patients will be asked to refrain from taking any medication or supplement to relieve their constipation.

After 14 days the patients will return and eligibility will be re-assessed. Patients will be trained on how to use the base unit.

Patients will be instructed to complete a simple patient eDiary each day throughout the duration of the study. After 3 weeks of treatment, the patient will attend for evaluation and to receive new capsules. A final visit will take place at the end of the 6 week treatment period.

Patients will receive phone calls up to twice per week and patient compliance will be monitored during the 8 weeks of the study.

ELIGIBILITY:
Inclusion criteria

1. Patients aged 22 years and older
2. Patients with Chronic Idiopathic Constipation according to Rome III criteria and who have not experienced relief of their symptoms from available therapies (osmotic and stimulant laxatives used for at least one month at recommended dose)
3. Patients with an average of less than 3 Spontaneous Bowel Movements per week and at least 1 Spontaneous Bowel Movements per week
4. Normal colonoscopy performed within 10 years prior to study participation, unless the patients are less than 50 years old and without alarm signs and/or symptoms
5. Patient signed the Informed Consent Form
6. Female subjects must have a negative urine pregnancy test and must not be lactating prior to receiving study medication. For females of child-bearing potential, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. All other female subjects must have the reason for their inability to bear children documented in the medical record; in these circumstances, a urine pregnancy test will not be necessary.

Exclusion criteria

1. History of complicated/obstructive diverticular disease
2. History of intestinal or colonic obstruction, or suspected intestinal obstruction.
3. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission)
4. History of gastroparesis
5. Use of any of the following medications:

   * Medications that may affect intestinal motility, prokinetics, anti-depressants, anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, aluminum/magnesium hydroxide
   * With the exception of antidepressants, thyroid or hormonal replacement therapy, when the subject has been on a stable dose for at least 3 months prior to enrollment.
6. Clinical evidence of significant respiratory, cardiovascular, renal, hepatic, biliary, endocrine, psychiatric or neurologic disease.
7. Presence of cardiac pacemaker or gastric electrical stimulator.
8. History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.
9. Diagnosis of mega-rectum or colon, congenital anorectal malformation, clinically significant rectocele, history of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit
10. History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia
11. Chronic use of non-steroidal anti-inflammatory drugs: chronic use is defined as taking full dose non-steroidal anti-inflammatory drugs more than three times a week for at least six months. Patients on cardiac doses of aspirin may be enrolled in the study
12. Patients with pelvic floor dysfunction/defecatory disorder, based on patient history
13. Participation in another clinical study within one month prior to screening.
14. Women who are pregnant or lactating
15. Use of any medication for constipation relief during the study, except as rescue medication, as indicated by study rules
16. Inability to use an electronic daily Diary (on a computer, phone application, tablet or other electronic device) to report bowel movements, symptoms and medication usage
17. Any other condition which in the opinion of the investigator may adversely affect the safety of the patient or would limit the patient's ability to complete the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eamonn Quigley, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (4):
- United States (4):
  - Avant Guntersville, Guntersville, Alabama
  - Borland-Groover Clinic, Jacksonville, Florida
  - Floridian Research Institute, Miami, Florida
  - Albuquerque Neuroscience, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No
Data from this study will be published in Vibrant's future publications

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vibrating Capsule
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vibrating Capsule
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Cacucasian | 3
  Hispanic or Latino | 21
  Native American or American Indian | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
Duration of constipation (years) [Mean (Standard Deviation); unit: years] | 12.2 (11.18)

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Bowel Movements Success Rate
Description: Defined as the number of subjects with an increase from the run-in period of at least one weekly Spontaneous Bowel Movement (SBM) during at least 3 of the 6 weeks of treatment. Subjects with less than 2 weeks (with at least 5 days per week) of valid diary during the treatment period will be considered as non-evaluable.
Time Frame: 6 weeks of treatment
Population: subjects with an improvement of at least 1 SBM a week, 3 out of 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrating Capsule
Number analyzed (Participants) | 24
Participants | 21

ADVERSE EVENTS:
Time Frame: For each patient, safety data was collected for 8 weeks of study participation.
Arm/Group | Vibrating Capsule
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vibrating Capsule (N=25)
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Emesis (Gastrointestinal disorders) | 1
exacerbation of kidney stones (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Permission to use study data is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT02829047/Prot_SAP_000.pdf